CLINICAL TRIAL: NCT03728660
Title: Design and Clinical Evaluation of a Smartphone-based Low Vision Enhancement System
Acronym: eLVES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Eye Institute (NEI) (NIH); Visionize, LLC (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB00086366; 4R44EY028077-02 (NIH)
Record Dates: First submitted 2018-10-31; First posted 2018-11-02 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2020-12

CONDITIONS: Low Vision
Keywords: age related macular degeneration; visual impairment; virtual reality
MeSH Terms: conditions — Vision, Low; Macular Degeneration; Vision Disorders

STUDY DESIGN:
Intervention Model Description: Intention to treat design; crossover with 22 week washout period between interventions; primary outcome measure is patient-reported function
Who Masked: Outcomes Assessor
Masking Description: Baseline AI administered prior to randomization, outcomes assessor masked on intervention assignment before and after crossover
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- LVES 2 first LEGACY second (Experimental): Virtual bioptic magnification with large field of view (LVES 2) followed by 22-week washout period and then Full field magnification with small field of view (LEGACY)
  Interventions: Device: Virtual bioptic magnification with large field of view; Device: Full field magnification with small field of view
- LEGACY first LVES 2 second (Active Comparator): Full field magnification with small field of view (LEGACY) followed by 22-week washout period and then Virtual bioptic magnification with large field of view (LVES 2)
  Interventions: Device: Virtual bioptic magnification with large field of view; Device: Full field magnification with small field of view

INTERVENTIONS:
Device: Virtual bioptic magnification with large field of view — The intervention device will have a larger field of vision than the legacy device and the intervention device will also have a virtual bioptic telescope mode not found on the legacy device. The user will be able to adjust the size of the virtual bioptic telescope and the amount of magnification with a touch pad on the side of the head-mounted display (HMD).
  Other Names: LVES 2; IrisVision
Device: Full field magnification with small field of view — Comparison intervention with user-controlled full field magnification with a smaller field size shared by legacy head-mounted devices. User can control amount of magnification
  Other Names: LEGACY

SUMMARY:
The primary objective is to compare the effectiveness and adverse side-effects of the virtual bioptic telescope and virtual projection screen in a new head-mounted video-based low vision enhancement system (LVES) with a wide field of view to currently employed specifications for head-mounted video display low vision enhancement technology. Secondary objectives are to acquire qualitative information from patients to evaluate the functioning of the system, to optimize system features and operations, and to assess the value patients place on system features, functions, and operating parameters relative to those of current technology. Investigators will conduct a comparative effectiveness study to determine if the novel vision enhancing features of LVES 2 provide low vision patients with benefits superior to those provided by existing technology.

DETAILED DESCRIPTION:
The study will employ a single center, randomized crossover design with a 2-week trial period before the crossover, a 22-week washout period, and a 2-week trial period after the cross over. Once recruited patients have consented to participate in eligibility screening for the study, participants will be administered the Activity Inventory (AI), a rating scale questionnaire about the difficulty of performing a wide range of daily activities and the Telephone Interview for Cognitive Status (TICS) Eligible patients who consent to participate will be randomized to Group A or Group B. Group A will be trained to use and will employ at home for the first 2-week trial period, the headset with the new LVES 2 features and specifications and then, after the 22-week washout period, will be trained to use and employ at home for the second 2-week trial period the headset with currently available features and specifications ("legacy system"). The order will be reversed for Group B who will start with the legacy system for trial period 1 and then switch to the new LVES 2 system for trial period 2 after the 22-week washout.

Prior to each 2-week trial period, participants will visit the laboratory and will be taught how to operate the new LVES 2. Once the participant is familiar with the basic control operations, he/she will receive one on one instruction from a low vision rehabilitation therapist on the use of the device with the features and specifications to be tested to perform distance, intermediate and near activities. Prior to dispensing either device for a 2-week home trial evaluation, the patient must demonstrate to the satisfaction of the therapist a basic knowledge of and successful operational skill with the device, including an understanding that participants are not to attempt to walk or operate a vehicle while wearing the device.

Guided by the AI results, participants will be instructed on the types of activities participants should perform at home while using the device. The participant will also take part in baseline testing in 1. Facial recognition, 2.Visual motor test, 3. The International Reading Speed Texts (IReST) to assess reading performance, and 4. a modified Timed Activity of Daily Living (TIADL) performance test. The patient will be called during the 2-week home trial period and a Simulator Sickness Questionnaire (SSQ) will be administered. A follow-up AI will be administered at the end of the 2-week trial. The participant will return the headset to the laboratory after the 2-week trial and will be debriefed on participant's experiences and impressions. The 4 tests will be repeated at this visit (Facial recognition, Visual motor, IReST and TIADL). None of these procedures are part of or substitute for the patient's routine care. Investigators will employ rolling enrollment of participants on staggered schedules. Investigators expect to complete the 50th participant with the first condition in 22 weeks and then Investigators will start the crossover phase after the 22-week washout. Investigators expect to complete both phases with the first 50 patients (less drop outs) in year 1. Investigators then repeat the procedure with the next group of 50 participants in year 2, using systems that include new software features developed in response to participant feedback.

A treatment success is defined as an improvement in functional ability measured with the Activity Inventory that exceeds the 95% confidence interval of the estimated baseline measure [i.e.,Minimum Clinically Important Difference (MCID)]. Stopping the home trial will not be initiated by the investigators, but participants who are experiencing significant simulator sickness will be encouraged to stop.

Participants who stop the home trial prematurely will still be asked to complete the post-trial debriefing and the follow-up AI. Since study participation does not substitute for the patient's regular clinical care, there is no consequence to the patient for prematurely ending study participation.

ELIGIBILITY:
Inclusion Criteria:

* Visual acuity in the better-seeing eye 20/60-20/800
* Horizontal visual field extent >70 degrees diameter, vertical visual field extent >50 degrees.
* Indicate at least 2 goals from the Activity Inventory during the initial screening interview.
* Scores at least 27 in the Telephone Interview Cognitive Status during the initial screening interview

Exclusion Criteria:

* Patients who are planning ocular surgery (including laser surgery) during the period of study participation or are early in anti-neovascular treatment (<6 injections)
* Younger than 14 years of age
* Unable to participate in a telephone interview
* Indicate less than 2 goals from the Activity Inventory
* Score less than 27 in the Telephone Interview Cognitive Status

Ages: 14 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2019-01-29 (Actual); Primary Completion 2021-02-05 (Actual); Study Completion 2021-02-05 (Actual)

PRIMARY OUTCOMES:
Mean change in patients' self-reported functional ability as assessed by the Activity Inventory (AI) rating scale questionnaire | 2 weeks, 24 weeks
  Functional ability is estimated from difficulty ratings of items in the AI, a questionnaire that banks 510 items describing common activities. 50 items are "goals", broad descriptions of activity accomplishments. The other 460 items are "tasks", specific activities typically performed to achieve goals. The patient rates the importance of each goal. Unimportant goals are skipped, otherwise the patient rates the goal's difficulty. If "not difficult", the patient skips to the next goal, otherwise rates the difficulty of the goal's subsidiary tasks, or responds "not applicable". The average ability required by each item and the functional ability of each patient are estimated on the same scale with Rasch analysis. The 510 item measures in the AI are fixed to values for 3000 low vision patients. The investigators will analyze functional ability change score distributions for the two interventions before and after the crossover.

SECONDARY OUTCOMES:
Minimum Clinically Important Difference (MCID) in patient's self-reported functional ability estimated from difficulty ratings of activities in the AI rating scale questionnaire | 2 weeks, 24 weeks
  MCID is a clinical endpoint defined as a change (an improvement) in the person measure from pre-trial period to post-trial period estimated from all items in the Activity Inventory identified by the patient as relevant and at least somewhat difficult at baseline that exceeds that patient's 95% confidence interval for person measure change (see the Outcome 1 description for details). MCID counts are repeated for the crossover after a 22-week washout period. The investigators will compare the rates of achieving MCID endpoints for the two intervention arms both before and after the crossover.

CONTACTS AND LOCATIONS:
Overall Officials: Robert W Massof, Ph.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
If individual participant data (IPD) is shared, it will be in the form of a csv data file included as supplemental material attached to the published results.

REFERENCES:
- [Background] Deemer AD, Bradley CK, Ross NC, Natale DM, Itthipanichpong R, Werblin FS, Massof RW. Low Vision Enhancement with Head-mounted Video Display Systems: Are We There Yet? Optom Vis Sci. 2018 Sep;95(9):694-703. doi: 10.1097/OPX.0000000000001278. PMID 30153240
- [Background] Goldstein JE, Jackson ML, Fox SM, Deremeik JT, Massof RW; Low Vision Research Network Study Group. Clinically Meaningful Rehabilitation Outcomes of Low Vision Patients Served by Outpatient Clinical Centers. JAMA Ophthalmol. 2015 Jul;133(7):762-9. doi: 10.1001/jamaophthalmol.2015.0693. PMID 25856370
- [Background] Massof RW, Ahmadian L, Grover LL, Deremeik JT, Goldstein JE, Rainey C, Epstein C, Barnett GD. The Activity Inventory: an adaptive visual function questionnaire. Optom Vis Sci. 2007 Aug;84(8):763-74. doi: 10.1097/OPX.0b013e3181339efd. PMID 17700339
- [Derived] Chun R, Deemer A, Fujiwara K, Deremeik J, Bradley CK, Massof RW, Werblin FS. Comparative effectiveness between two types of head-mounted magnification modes using a smartphone-based virtual display. Optom Vis Sci. 2024 Jun 1;101(6):342-350. doi: 10.1097/OPX.0000000000002115. Epub 2024 Apr 12. PMID 38551973